CLINICAL TRIAL: NCT02440542
Title: Popliteal Nerve Block for Postoperative Pain Control in Patients Undergoing Ankle and Hindfoot Reconstruction About the Talus
Brief Title: Popliteal Nerve Block for Postoperative Pain Control in Ankle and Hindfoot Reconstruction
Status: Withdrawn | Type: Observational
Why Stopped: Study enrollment not initiated due to institutional delays
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Other Study IDs: 15-025
Record Dates: First submitted 2015-04-20; First posted 2015-05-12 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Pain, Postoperative
Keywords: Nerve block; Ankle; Talus; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Postoperative Popliteal nerve block: All patients in the cohort are receiving a postoperative popliteal nerve block as part of their surgical plan. Outcomes including length of stay, Visual Analog Scale Scores, narcotic intake, and patient satisfaction will be collected as the intervention.
  Interventions: Other: Survey of outcomes following popliteal nerve block

INTERVENTIONS:
Other: Survey of outcomes following popliteal nerve block — Patients will be instructed to complete journals of pain and narcotic use until postoperative day 10. On first follow-up visit, patients will complete a patient satisfaction survey. VAS Pain scores and pain medication use will be collected up to 12 weeks postoperatively.

SUMMARY:
The purpose of this study is to evaluate outcomes of popliteal nerve blocks for postoperative pain control in patients undergoing ankle and hindfoot reconstruction surgeries. The following outcomes will be analyzed: length of hospital stay, level of pain control, pain medication use, complications, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years old
* Patients undergoing ankle, subtalar, pantalar, triple, or tibiotalocalcaneal arthrodesis (CPT codes 27870, 28715, 28725, or 28740)
* Patients undergoing total ankle arthroplasty (CPT code 27702)
* Patients with a preoperative surgical plan to receive a popliteal nerve block during the postoperative period
* Patients whom can be reasonably expected to understand and comply with patient-reported postoperative data collection and surveys

Exclusion Criteria:

* Patients undergoing an ankle or hindfoot reconstruction procedure whom are medically ineligible to receive a safe popliteal nerve block (i.e. patients with neuropathy)
* Patients with documented substance abuse (i.e. history of narcotic abuse could confound pain outcomes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be patients undergoing ankle or hindfoot reconstruction about the talus (ankle arthrodesis, subtalar arthrodesis, or ankle arthroplasty) who will be receiving a sciatic nerve block in the popliteal region while in the PACU, following surgery. Patients will be identified as potential subjects from within the practices of two fellowship-trained foot and ankle orthopaedic surgeons. Patients will be enrolled in the study by Informed Consent
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Pain rating | Postoperative- through 12 weeks
  Measured by VAS

SECONDARY OUTCOMES:
Narcotic intake | Postoperative- through 12 weeks
  Measured by data from hospital medical record and patient questionnaire
Hospital length of stay | Postoperative- through day of hospital discharge (discharge same day of surgery to approximately 3 days postop)
  Measured by data from hospital medical record
Patient satisfaction | Postoperative- through first surgical follow-up (up to 3 weeks)
  Measured by patient questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jesse F Doty, MD, Principal Investigator — University of Tennessee College of Medicine Chattanooga/Erlanger Health System